CLINICAL TRIAL: NCT02652871
Title: A Phase 1b, Open-label Study of LY2510924, Idarubicin and Cytarabine in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: LY2510924, Idarubicin and Cytarabine in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry); High Impact Clinical Research Support Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0436; NCI-2016-00259 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Leukemia
Keywords: Leukemia; Acute Myeloid Leukemia; AML; Relapsed or Refractory; Acute myelogenous leukemia; LY2510924; Idarubicin; Idamycin; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Recurrence | interventions — LY2510924; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY2510924 + Idarubicin + Cytarabine (Experimental): Dose Escalation Phase: Starting dose level of LY2510924 is 10 mg subcutaneously each day of a 28 day cycle. Dose escalated in successive cohorts of patients. On Day 8, LY2510924 administered after bone marrow aspiration and/or biopsy is performed.
  Dose Expansion Phase: LY2510924 given at the maximum tolerated dose (MTD) from Dose Escalation Phase.
  Dose Escalation Phase: Idarubicin 12 mg/m2 by vein given on Days 8 and 9 of a 28 day cycle. In patients > 60 years of age Idarubicin given for 2 days.
  Dose Expansion Phase: Idarubicin 8 mg/m2 by vein for 2 days.
  Dose Escalation Phase: Cytarabine 1.5 gm/m2 by vein daily for 4 days (age < 60 years). In patients > 60 years of age Cytarabine given for 3 days only.
  Dose Expansion Phase: Cytarabine 0.75 gm/m2 by vein for 3 days.
  Interventions: Drug: LY2510924; Drug: Idarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: LY2510924 — Dose Escalation Phase: Starting dose level of LY2510924 is 10 mg subcutaneously each day of a 28 day cycle. Dose escalated in successive cohorts of patients.
  Dose Expansion Phase: LY2510924 given at the maximum tolerated dose (MTD) from Dose Escalation Phase.
Drug: Idarubicin — Dose Escalation Phase: Idarubicin 12 mg/m2 by vein given on Days 8 and 9 of a 28 day cycle. In patients > 60 years of age Idarubicin given for 2 days.
  Dose Expansion Phase: Idarubicin 8 mg/m2 by vein for 2 days.
  Other Names: Idamycin
Drug: Cytarabine — Dose Escalation Phase: Cytarabine 1.5 gm/m2 by vein daily for 4 days (age < 60 years). In patients > 60 years of age Cytarabine given for 3 days only.
  Dose Expansion Phase: Cytarabine 0.75 gm/m2 by vein for 3 days.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride

SUMMARY:
The goal of this clinical research study is to learn about the safety of LY2510924 in combination with cytarabine and idarubicin in patients with relapsed or refractory AML. We will also study if LY2510924 in combination with cytarabine and idarubicin can help to control relapsed or refractory AML.

LY2510924 is designed to help cancer cells move from the bone marrow into the bloodstream, where they are exposed to chemotherapy (in this case, cytarabine and idarubicin).

This is an investigational study. LY2510924 is not FDA approved or commercially available. Its use in this study is investigational. Cytarabine and idarubicin are approved to treat certain types of leukemia. Their use in this study in combination with LY2510924 is investigational.

Up to 36 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 3 groups of up to 6 participants each will be enrolled in the Dose Escalation part of the study, and up to 18 participants will be enrolled in Dose Expansion part of the study.

If you are enrolled in the Dose Escalation part of the study, the dose of LY2510924 you receive will depend on when you join this study. The first group of participants will receive the lowest dose level of LY2510924. Each new group will receive a higher dose of LY2510924 than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of LY2510924 is found.

If you are enrolled in the Dose Expansion part of the study, you will receive LY2510924 at the highest dose that was tolerated in the Dose Expansion part of the study.

All participants will also receive idarubicin and cytarabine. Your dose level will be assigned based on your age.

Study Drug Administration:

Treatment on this study is given in 2 phases: Induction and Consolidation. Each phase is made up of 28-day study cycles.

Induction Phase:

You will receive 1-2 cycles during the Induction phase. During Cycle 1, you will be admitted to the inpatient Leukemia service when you receive the study drugs.

You will receive LY2510924 alone each day for 7 days and then together with chemotherapy on Days 8, 9 and 10 and also on Day 11 if you are under the age of 60, of every 28-day cycle.

* On days that you do not receive idarubicin/cytarabine, LY2510924 will be given as an injection under the skin at about 8:00 am (+/- 1½ hours).
* On days when you do receive idarubicin/cytarabine, it will be given about 4 hours (+/- ½ hour) before you receive idarubicin.

On Days 8 and 9, in addition to LY2510924:

* You will receive idarubicin by vein over about 1 hour.
* You will receive cytarabine by vein over about 24 hours.

On Day 10, in addition to LY2510924:

* You will receive cytarabine by vein over about 24 hours.
* If you are under age 60, you will receive idarubicin by vein over about 1 hour.

If you are under age 60, on Day 11, in addition to LY2510924, you will receive cytarabine by vein over about 24 hours.

On days that you are receiving the cytarabine infusions, you will receive drugs to help reduce the risk of side effects. You will receive dexamethasone before the cytarabine infusion by vein over about 30 minutes. You will also receive corticosteroid-containing eye drops during this time and for 2 days following the last dose of cytarabine.

If the disease does not respond during Cycle 1, you may be allowed to receive an additional Induction cycle, which will also be called Cycle 1.If you do respond to Induction, you can move to the Consolidation phase.

Consolidation Phase:

If you are benefitting from the treatment, you may continue with Consolidation therapy for an additional 4-6 cycles.

During these cycles, you will receive LY2510924 in the same way as during earlier cycles, for 3 days with chemotherapy. During Consolidation, all participants will receive idarubicin by vein over 1 hour on Days 1 and 2, and cytarabine by vein over 24 hours on Days 1-3.

Study Visits:

During Days 1-12 of Cycle 1 (if over the age of 60, Days 1-10), blood (about 4 teaspoons) will be drawn for routine tests. During Days 1-7, blood (about 2 teaspoons) will be drawn 4 hours after your injection with LY2510924 for routine tests.

On Days 8 and 28 of Cycle 1, you will have a bone marrow biopsy/aspirate to check the status of the disease.

After Day 11 of Cycle 1, blood (about 4 teaspoons) will be drawn every 2-4 days for routine tests.

Every 1-2 weeks during Cycles 2-6, blood (about 4 teaspoons) will be drawn for routine tests.

Every 2-4 weeks during Cycles 2-6, you will have a physical exam.

After Cycles 4 and 6, you will have a bone marrow biopsy and aspiration to check the status of the disease. You will also have an EKG and either an ECHO or MUGA scan.

Any time the doctor thinks it is needed, you will have additional blood tests.

Length of Study:

You may receive up to 8 cycles of the study drugs. You will be taken off study if the disease gets worse, you experience intolerable side effects, or if the study doctor thinks it is in your best interest.

Your participation on this study will be over after you complete the End-of-Treatment Visit.

End-of-Treatment Visit:

About 30 days (+/- 5 days) after your last dose of the study drugs, blood (about 2 teaspoons) will be drawn for routine tests.

Long Term Follow-up:

Every 2-3 months for up to 2 years after you stop receiving the study drugs, blood (about 4 teaspoons) will be drawn for routine tests. This can be performed at your local doctor's office. You should also have a bone marrow aspiration/biopsy every 3 months for the first year, and then more after that if the doctor thinks it is in your best interest. If any of these tests show abnormal results, you will return to the study clinic for follow-up testing.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with histologically or cytologically confirmed relapsed or refractory AML [except acute promyelocytic leukemia]; relapsed disease or refractory (refractory to a non-high-dose cytarabine-containing regimen only); receiving 1st, 2nd or 3rd salvage; any cytogenetic or molecular abnormality. Patients with secondary AML (after prior myelodysplasia or therapy for other cancers) will be included.
2. Patients with prior autologous and allogeneic hematopoietic stem cell transplantation are eligible if patients are off immunosuppression for greater than 14 days and have no evidence of active graft versus host disease (GVHD) except grade 1 skin GVHD.
3. Clinical laboratory values should be as follows: (a) White blood count < 30,000/µL; (b) Absolute Blasts in peripheral blood < 20,000 (treatment with Hydroxyurea is permitted up to 24 hrs prior to LY251092 administration to achieve blast counts < 20,000 prior to enrollment).
4. Patients must be 18-70 years old.
5. Patients must have a performance status of 0-2 (Zubrod scale).
6. Patients must have adequate renal function (serum creatinine less than or equal to 1.3 mg/dL). If creatinine is > 1 mg/dL the creatinine clearance should be > 40 mL/min as calculated using the Cockcroft-Gault formula.
7. Patients must have adequate hepatic function (bilirubin less than or equal to 2.0 mg/dl; serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) less than or equal to 3 X the upper limit of normal [ULN] for the reference lab unless due to leukemia or congenital hemolytic disorder or bilirubin excretion disorder). Patients with hepatic dysfunction (SGOT/SGPT up to less than or equal to 5 X ULN) due to organ infiltration by disease may be eligible after discussion with the Principal Investigator and appropriate dose adjustments will be considered.
8. Patients must have normal cardiac ejection fraction (left ventricular ejection fraction [LVEF] greater than or equal to 50%).
9. Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study, in keeping with the policies of the hospital.
10. Negative urine or blood pregnancy test for women of childbearing potential.
11. Female patients must not be pregnant or lactating. Female patients of childbearing potential (including those <1 year post-menopausal) and male patients must agree to use contraception.

Exclusion Criteria:

1. Patients with untreated or uncontrolled life-threatening infection.
2. Patients who have received chemotherapy and/or radiation therapy within 2 weeks unless there is evidence of rapidly progressive disease. In the event that subjects have received chemotherapy < 2 weeks from the date of enrollment, they may be included provided they have recovered from the associated non-hematological toxicities to less than or equal to grade 1. Hydroxyurea is allowed up to 24 hours prior to starting therapy in the setting of rapidly proliferating disease.
3. Patients who have received an investigational anti-cancer drug within two weeks (or five half-lives, whichever is shorter) of LY251092 administration.
4. History of myocardial infarction or cerebrovascular accident within 6 months of enrollment date.
5. History of another malignancy. Exception: Patients who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies, are eligible.
6. Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent or cooperate and participate in the study or with the interpretation of the results.
7. Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression (patients with controlled central nervous system (CNS) disease, i.e. asymptomatic and currently receiving concurrent intrathecal chemotherapy, are eligible upon discussion with the Principal InvestigatorI).
8. Known active Hepatitis B Virus (HBV), Human Immunodeficiency Virus (HIV) or Hepatitis C Virus (HCV) infection (patients with chronic or cleared HBV and HCV infection, are eligible).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-05-09 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity of LY2510924, Idarubicin and Cytarabine in Patients with Relapsed or Refractory Acute Myeloid Leukemia | 30 days post transplant
  Dose-limiting toxicity (DLT) defined as a clinically significant adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness or concomitant medications. To be considered a DLT such toxicity must be possibly, probably or definitely related to LY2510924. Toxicity evaluated using the National Cancer Institute (NCI) Version 4.0 criteria.

SECONDARY OUTCOMES:
Response of LY2510924, Idarubicin and Cytarabine in Patients with Relapsed or Refractory Acute Myeloid Leukemia | 56 days
  International Working Group Criteria used to define response.
  Complete remission (CR): Participant must be free of all symptoms related to leukemia and have an absolute neutrophil count (ANC), 1.0 x 109/L, platelet count, 100 x 109/L, and normal bone marrow differential (5% blasts).
  Complete remission without platelet recovery (CRp): As per CR but platelet count 100 x 109/L.
  Complete Remission with Incomplete Blood Count Recovery (CRi): Peripheral blood and bone marrow results as for CR except for ANC < 1.0 x 109/L with or without platelet count < 100 x 109/L.
  Partial remission (PR): CR with 6 to 25% abnormal cells in the marrow or 50% decrease in bone marrow blasts.
  Morphologic leukemia-free state: Normal marrow differential (5% blasts); neutrophil and platelet counts are not considered.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Konopleva, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org